CLINICAL TRIAL: NCT05573763
Title: Evaluation of the F&P Toffee Nasal Pillows Mask, US, 2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-308
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- single-arm, non-randomized, and open-label (Other)
  Interventions: Device: F&P Toffee

INTERVENTIONS:
Device: F&P Toffee — Nasal pillows mask

SUMMARY:
The purpose of this clinical investigation is to evaluate the performance and safety of the F&P Toffee nasal pillows mask in a home environment.

ELIGIBILITY:
Inclusion Criteria:

* Persons who are ≥22 years of age
* Persons who weigh ≥66 pounds
* Persons who have been prescribed PAP therapy by a physician
* Persons who are existing nasal pillows mask users with at ≥3 months of use prior to enrolment in the clinical trial
* Persons who are compliant with PAP therapy for ≥4 hours per night for ≥70% of nights for a 14-day period within 30 days prior to enrolment in the clinical trial
* Persons who are fluent in spoken and written English
* Persons who possess the capacity to provide informed consent

Exclusion Criteria:

* Persons who are intolerant to PAP therapy
* Persons who possess, or suffer from, anatomical or physiological conditions which make PAP therapy inappropriate
* Persons who are required to use PAP therapy for >12 hours per day or for extensive periods, not including sleep or naps
* Persons who are trying to get pregnant, are pregnant, or think they may be pregnant
* Persons who have an IPAP pressure of >25 cmH2O if on BPAP
* Persons who use a PAP therapy device for the delivery of medicines, except supplemental O2
* Persons who use a PAP therapy device that does not possess data recording capabilities to capture AHI and a numerical indicator of leak that is accessible to the investigation site

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio Sleep Medicine Institute, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Toffee: Nasal Pillows Mask: Participants to use nasal pillows mask for 14 days. Nasal Pillows Mask: Nasal Pillows mask for the treatment of obstructive sleep apnea (OSA)
Period: Overall Study
Arm/Group | Toffee: Nasal Pillows Mask
Started | 40
Completed | 39
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- F&P Toffee: Nasal Pillows Mask: Participants to use nasal pillows mask for 14 days. Toffee Nasal Pillows Mask: Nasal Pillows mask for the treatment of obstructive sleep apnea (OSA)
Arm/Group | F&P Toffee: Nasal Pillows Mask
Number analyzed (Participants) | 39
Age, Customized [Count of Participants; unit: Participants]
  22+ years of age | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Efficacy
Description: Determined by Apnea-Hypopnea Index (AHI) recorded on PAP therapy machines after 14 days of use. The Apnea-Hypopnea index (AHI) is the sum of the apneas and hypopneas divided by the hours of sleep. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and >= 30/h = severe"
Time Frame: Baseline and 14±5 days
Measure: Mean (Full Range); unit: events per hour
Groups:
- F&P Toffee: Nasal Pillows Mask: Participants will be placed in the experimental arm for 14 days, during which they will be using either the Toffee Nasal or Toffee Nasal Pillows mask for PAP therapy.
  F&P Toffee Nasal and Toffee Nasal Pillows Masks: F&P Toffee Nasal and Toffee Nasal Pillows Masks are intended to be used within the traditional PAP therapy system and are designed to facilitate equivalent PAP therapeutic efficacy as defined by standard practice.
Arm/Group | F&P Toffee: Nasal Pillows Mask
Number analyzed (Participants) | 39
events per hour | 2 [0.3 to 4.5]

2. Primary Outcome: Epworth Sleepiness Scale
Description: All relevant time points used in the calculation in the Time Frame (e.g., baseline and 14±5 days).
  Note: change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 14±5 days minus value at baseline).
  Change between two time points is reported. Scale range: 0 (minimum score) to 24 (maximum score) (higher scores represent worse outcomes)
Time Frame: 14±5 days
Measure: Mean (Full Range); unit: Scores on a scale
Groups:
- Toffee: Nasal Pillows Mask: Participants to use nasal pillows mask for 14 days. Toffee Nasal Pillows Mask: Nasal Pillows mask for the treatment of obstructive sleep apnea (OSA)
Arm/Group | Toffee: Nasal Pillows Mask
Number analyzed (Participants) | 39
Scores on a scale | 10 [0 to 13]

ADVERSE EVENTS:
Time Frame: 14 days
Description: 0
Arm/Group | F&P Toffee: Nasal Pillows Mask
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 2/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F&P Toffee: Nasal Pillows Mask (N=39)
Sinus Cold (General disorders) | 1 (1) — sinus cold/infection
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1) — Shoulder and back pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT05573763/Prot_SAP_002.pdf